CLINICAL TRIAL: NCT06670482
Title: The Effect of Mask Design on Transcutaneous Carbon Dioxide in Healthy Volunteers: A Pilot Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIA-351; U1111-1313-6217 (Other: World Health Organisation)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers; Noninvasive Ventilation
Keywords: Non-invasive ventilation; mask; Transcutaneous CO2
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, non-blinded
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): NIV using Mask A, with mouth-open
  Interventions: Device: Non-invasive ventilation (NIV)
- Arm 2 (Experimental): NIV using Mask A, with mouth-closed
  Interventions: Device: Non-invasive ventilation (NIV)
- Arm 3 (Active Comparator): NIV using Mask B, with mouth-open
  Interventions: Device: Non-invasive ventilation (NIV)
- Arm 4 (Active Comparator): NIV using Mask B, with mouth-closed
  Interventions: Device: Non-invasive ventilation (NIV)

INTERVENTIONS:
Device: Non-invasive ventilation (NIV) — Delivery of positive airway pressure to the lungs via an interface, such as a mask.

SUMMARY:
The goal of this randomized cross-over study is to investigate whether the design of non-invasive ventilation (NIV) mask impacts transcutaneous CO2 in healthy volunteers on NIV therapy. The main questions it aims to answer are:

* To assess if mask design impacts transcutaneous CO2 in healthy volunteers.
* To assess if mask design impacts tidal volume or respiratory rate in healthy volunteers.

Participants will attend three study visits:

* Visit 1. Participants will be fitted to use non-invasive ventilation briefly to acclimatize them to using the therapy.
* Visit 2. Participants will receive NIV with one of two masks. They will be asked to breathe through their mouth or through their nose, with a break from NIV in between the two sessions of NIV.
* Visit 3. Participants will receive NIV with the other mask, repeating Visit 2.

DETAILED DESCRIPTION:
The study compares breathing with two different NIV masks, the interventional mask and the conventional NIV mask. Participants will be monitored by transcutaneous carbon dioxide, electrical impedance tomography (EIT) and heart rate, oxygen and respiratory rate monitors.

Participants will attend three study visits:

* Visit 1. Participants will be fitted to use NIV briefly to acclimatize them to using the therapy and ensure the two study masks fit. Participants that fit the masks and tolerate NIV well will be invited to attend two further visits.
* Visit 2. Participants will be randomized as to which order they receive the masks and which order they conduct mouth breathing and nose breathing. Baseline readings of normal unsupported breathing will be taken prior to going on NIV. Participants will the receive NIV with one of two masks for ten minutes, and will be instructed to either breathe with their mouth open or their mouth closed. There will then be a break from NIV of at least ten minutes until baseline values of respiratory parameters have returned. Then there will be a second ten minute period of NIV when the participant will be instructed to breathe through the other way - mouth-closed or mouth-open. One NIV therapy has been removed the participant will remain attached to the study monitoring equipment until respiratory parameters have returned to normal.
* Visit 3 is a repeat of Visit 2 with the other study mask. The study is then complete.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Able to give informed consent

Exclusion Criteria:

* Unable to tolerate non-invasive ventilation (NIV)
* Unable to adequately fit an NIV mask
* Claustrophobia while using NIV
* Reported pregnancy
* Symptoms of cold or flu (included COVID-19) in previous twenty four hours
* Pneumothorax or history of previous pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Change in transcutaneous carbon dioxide (CO2) | Continuous assessment collected during baseline normal breathing and from the start to the finish of each NIV session.
  To assess if mask design can reduce transcutaneous CO2, in healthy volunteers.

SECONDARY OUTCOMES:
Change in respiratory rate | Continuous assessment collected during baseline normal breathing and from the start to the finish of each NIV session.
  To assess if mask design can reduce respiratory rate in healthy volunteers.
Change in tidal volume | Continuous assessment collected during baseline normal breathing and from the start to the finish of each NIV session.
  To assess if mask design can reduce tidal volume in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: William Good, MD, Principal Investigator — Middlemore Hospital, New Zealand
Locations (1):
- Fisher and Paykel Healthcare, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
All data to be deidentified.